CLINICAL TRIAL: NCT05140317
Title: 5 Years Hemodynamic and Clinical Follow-up of the SAPIEN 3 Transcatheter Heart Valve According to the Implantation Strategy: Insight From the Randomized DIRECTAVI Trial
Brief Title: 5 Years Follow up of the SAPIEN 3 Valve From the DIRECTAVI Trial
Acronym: DIRECTAVILONG
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0342
Record Dates: First submitted 2021-11-10; First posted 2021-12-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Coronary Syndrome; Hemodynamic Instability
Keywords: patients included in the directavi trial; TAVR Hemodynamic performances long term follow up
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: The direct stargegy group included patients with implanation of the THV without predilatation The reference group included patients with direct implanation of tne THV withour predilaation
  Interventions: Procedure: Transcatheter heart valve implantation with or withour predilatatation
- Group 2: the echographists were blinded regarding the groups of the patients
  Interventions: Procedure: Transcatheter heart valve implantation with or withour predilatatation

INTERVENTIONS:
Procedure: Transcatheter heart valve implantation with or withour predilatatation — long term up to 5 years echographic and clinical follow up

SUMMARY:
A strategy of Transcatheter Aortic Valve Replacement (TAVR) without balloon predilatation has shown to be feasible in routine in observational studies and in two recent randomized trial including the DIRECTAVI trial. Whether the initial implantation strategy may impact the long-term trans catheter heart valve (THV) performances and patient outcomes remains unknown to date. The Investigators therefore aimed to evaluate the 5-years impact of the implantation strategy on THV hemodynamic performances and clinical outcomes in patients included in the DIRECTAVI trial.

DETAILED DESCRIPTION:
All patients (n=236) included in the DIRECTAVI randomized trial conducted between May 2016 to May 2018 will be prospectively assessed for up to 5 years follow-up . The DIRECTAVI prospective, randomized, single-center, open-label trial, demonstrated the non-inferiority of a "direct TAVR" strategy using the third-generation balloon-expandable Edwards SAPIEN 3 device (Edwards Lifesciences, Irvine, CA, USA)

A systematic echographic follow-up will be performed in all patients enrolled in the DIRECTAVI trial at the longest follow -up obtained after TAVR between 2021 and 2022. Clinical follow-up will be obtained with a brief patient clinical questionnaire or by phone by patients' cardiologist.

Serial Echographic follow-up will be obtained by patients' cardiologist except for the latest follow-up echocardiography (primary end point) performed in the reference center at Montpellier University hospital by two experienced cardiologists specialized in valvular echography to avoid inter operator variability.

ELIGIBILITY:
Inclusion criteria:

* Older than 18 years old.
* patients included in the DIRECTAVI trial

Exclusion criteria:

- Patients not living in France

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients included in the DIRECTAVI trial
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
the incidence of patients without THV dysfunction | up to 5 years
  the incidence of patients without THV dysfunction according to the implantation strategy group (direct implantation vs ballon predilatation) at the latest follow-up available (up to 5 years)
the incidence of patients without correct hemodynamic performance | up to 5 years
  the incidence of patients without correct hemodynamic performance according to the implantation strategy group (direct implantation vs ballon predilatation) at the latest follow-up available (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Florence Leclercq, PU PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Jammoul N, Dupasquier V, Akodad M, Meunier PA, Moulis L, Soltani S, Macia JC, Robert P, Schmutz L, Steinecker M, Piot C, Targosz F, Benkemoun H, Lattuca B, Roubille F, Cayla G, Leclercq F. Long-term follow-up of balloon-expandable valves according to the implantation strategy: insight from the DIRECTAVI trial. Am Heart J. 2024 Apr;270:13-22. doi: 10.1016/j.ahj.2024.01.005. Epub 2024 Jan 20. PMID 38253304